CLINICAL TRIAL: NCT05827276
Title: Effects of the Life Story Questionnaire on Physical Therapy Participation in Patients With Dementia: A Randomized Control Trial
Brief Title: Life Story Questionnaire and Physical Therapy Participation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Texas Tech University Health Sciences Center (Other)
Collaborators: Texas Tech University (Other)
Responsible Party: Principal Investigator, Jean Michel Brismee, Principal co-investigator, Texas Tech University Health Sciences Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB2023-103
Record Dates: First submitted 2023-03-17; First posted 2023-04-25 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-04

CONDITIONS: Dementia Alzheimers
Keywords: Dementia; Life story questionnaire; Physical therapy; Physiotherapy; Participation; Exercise
MeSH Terms: conditions — Alzheimer Disease; Dementia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Control Trial. Patients will be randomly allocated in two groups: (1) Control group, which will receive standard physical therapy care without LSQ use; and (2) Experimental group, where physical therapists will use the LSQ.
Who Masked: Participant, Outcomes Assessor
Masking Description: The outcome assessor will be blind to the usage of the life story questionnaire for study participants. Additionally, the participants will not be told the group they were allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usage of Life Story Questionnaire (Experimental): This group will receive 6 weeks of physical therapy treatment as usual with the usage of the Life story questionnaire.
  Interventions: Other: Life story questionnaire
- No usage of Life Story Questionnaire (No Intervention): This group will receive 6 weeks of physical therapy treatment as usual with no usage of the Life Story Questionnaire.

INTERVENTIONS:
Other: Life story questionnaire — Participant will receive physical therapy treatment as usual using information from Life Story Questionnaire.
  Arms: Usage of Life Story Questionnaire

SUMMARY:
The goal of this clinical trial is to see the effect of life story questionnaire (LSQ) on physical therapy participation in patients with dementia. The main question[s] it aims to answer are:

1. What is the effect of LSQ usage on physical therapy participation in people with dementia?
2. What is the effect of LSQ usage on depression in people with dementia?
3. What is the effect of LSQ usage on the quality of life in people with dementia? The researcher will compare these effects between the intervention group (usage of the Life Story Questionnaire) and the control group (no usage of the Life story questionnaire).

All Participants will receive Physical therapy treatment as usual. The life Story Questionnaire will be used in the intervention group during physical therapy treatment.

Life Story Questionnaire: It is developed by the Crisis Prevention Institute, which is a type of life story book for people with dementia. The LSQ allows caregivers to start conversations about topics that are important to each patient, can help establish rapport between the caregiver and patient.

DETAILED DESCRIPTION:
Background: Dementia is characterized by a progressive decline in cognitive function. Dementia disease prevalence is substantially increased among people aged 65 years or older, with a progressive decline in memory, thinking, language and learning capacity. Although physical exercise benefits dementia patients, participation in activities is exceedingly difficult due to communication and cognitive impairments. Several studies demonstrated that life story books usage improved quality of life, depression symptoms, moods and participation in activity in people with dementia. However, these studies did not evaluate the effect of Life Story Questionnaire (LSQ) - a type of life story book - on physical therapy participation, depression symptoms, quality of life.

Objectives: To evaluate the impact of LSQ on (1) participation in physical therapy using Pittsburgh Rehabilitation Participation Scale; (2) quality of life using Quality of Life - Alzheimer's Disease Scale (participant's version); and (3) depression symptoms using Cornell Scale for Depression in Dementia (CSDD).

Methods: A consecutive sample of convenience of up to 60 patients with mild to moderate cognitive impairment with 44 (22 per group) completing the study will be recruited from a nursing home facility. Patients will be randomly allocated in two groups: (1) Control group, which will receive standard physical therapy care without LSQ use; and (2) Experimental group, where physical therapists will use the LSQ. Each patient's family member will receive a LSQ to complete prior to the start of the intervention. Patients' participation, quality of life and depression symptoms will be measured on day 1 and again after 3 weeks (mid-term), and 6 weeks of intervention. Quality of life and depression symptoms will also be measured 6 weeks following intervention. A licensed occupational therapist blinded to the participants' group allocation will measure all three dependent variables

Statistical Analysis: Descriptive statistics including means, standard deviations, frequency counts, median, mode, variance and frequency counts will be used to assess sample demographics. The Rank Sum test will be used to assess differences in Pittsburgh Rehabilitation Participation Scale between the intervention and control group. Spearman Rank correlations will be used to determine the strength of the correlation between Mini-Mental state examination, Pittsburgh Rehabilitation Participation Scale and Quality of Life Alzheimer Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients residing at dementia facility in Texas;
2. Age 60-89 years;
3. Diagnosis of dementia disease, in mild to the moderate stage using the Mini-Mental State Examination (score between 10 -24) and
4. Attendance to physical therapy for 6 weeks.

Exclusion Criteria:

1. Unable to speak English;
2. Blindness;
3. Deafness;
4. Mini-Mental State Examination score >24 and
5. history of major psychiatric disorders such as schizophrenia and bipolar disorder requiring hospital admission within the last year.

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Rehabilitation Participation Scale | 1st week of physical therapy
  To measure participation in physical therapy. Participation is graded as none (1), Poor (2), Fair (3), Good (4), Very good (5), and Excellent (6). Higher score indicates greater participation in physical therapy sessions.
Pittsburgh Rehabilitation Participation Scale | 3rd week of Physical Therapy
  To measure participation in physical therapy. Participation is graded as none (1), Poor (2), Fair (3), Good (4), Very good (5), and Excellent (6). Higher score indicates greater participation in physical therapy sessions.
Pittsburgh Rehabilitation Participation Scale | 6th week of Physical Therapy
  To measure participation in physical therapy. Participation is graded as none (1), Poor (2), Fair (3), Good (4), Very good (5), and Excellent (6). Higher score indicates greater participation in physical therapy sessions.

SECONDARY OUTCOMES:
Quality of life in Alzheimer's disease scale- participant's version | 1st week of Physical Therapy
  The quality of life in Alzheimer's disease scale rates 13 types of life domains and uses a scale of poor (1), fair (2), good (3), and excellent (4). Minimum score is 13 and maximum score is 52. Higher scores indicate better quality of life.
Quality of life in Alzheimer's disease scale- participant's version | 3rd week of Physical Therapy
  The quality of life in Alzheimer's disease scale rates 13 types of life domains and uses a scale of poor (1), fair (2), good (3), and excellent (4). Minimum score is 13 and maximum score is 52. Higher scores indicate better quality of life.
Quality of life in Alzheimer's disease scale- participant's version | 6th week of Physical Therapy
  The quality of life in Alzheimer's disease scale rates 13 types of life domains and uses a scale of poor (1), fair (2), good (3), and excellent (4). Minimum score is 13 and maximum score is 52. Higher scores indicate better quality of life.
Quality of life - Alzheimer's disease - participant's version | 6 weeks following intervention of Physical Therapy
  The quality of life in Alzheimer's disease scale rates 13 types of life domains and uses a scale of poor (1), fair (2), good (3), and excellent (4). Minimum score is 13 and maximum score is 52. Higher scores indicate better quality of life.

OTHER OUTCOMES:
Cornell scale for depression in dementia | 1st week of Physical Therapy
  It is a a screening tool and assesses depression symptoms in dementia participants. Score ranges from a - unable to evaluate, 0- absent, 1- mild, 2- severe. Minimum score is 0 and maximum score is 38. Higher scores indicate greater depression.
Cornell scale for depression in dementia | 3rd week of Physical Therapy
  It is a a screening tool and assesses depression symptoms in dementia participants. Score ranges from a - unable to evaluate, 0- absent, 1- mild, 2- severe. Minimum score is 0 and maximum score is 38. Higher scores indicate greater depression.
Cornell scale for depression in dementia | 6th week of Physical Therapy
  It is a a screening tool and assesses depression symptoms in dementia participants. Score ranges from a - unable to evaluate, 0- absent, 1- mild, 2- severe. Minimum score is 0 and maximum score is 38. Higher scores indicate greater depression.
Cornell scale for depression in dementia | 6 weeks following intervention of Physical Therapy
  It is a a screening tool and assesses depression symptoms in dementia participants. Score ranges from a - unable to evaluate, 0- absent, 1- mild, 2- severe. Minimum score is 0 and maximum score is 38. Higher scores indicate greater depression.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Brismee, ScD, Principal Investigator — Texas Tech University Health Sciences Center; Jonathan Singer, PhD, Principal Investigator — Texas Tech University
Locations (1):
- Peachtree Place (Dementia care facility), Weatherford, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 2018 Alzheimer's Disease Facts and figures" (2018) Alzheimer's & Dementia, 14(3), pp. 367-429. Available at: https://doi.org/10.1016/j.jalz.2018.02.001.
- [Background] Arvanitakis Z, Bennett DA. What Is Dementia? JAMA. 2019 Nov 5;322(17):1728. doi: 10.1001/jama.2019.11653. No abstract available. PMID 31688886
- [Background] Machiels M, Metzelthin SF, Hamers JP, Zwakhalen SM. Interventions to improve communication between people with dementia and nursing staff during daily nursing care: A systematic review. Int J Nurs Stud. 2017 Jan;66:37-46. doi: 10.1016/j.ijnurstu.2016.11.017. Epub 2016 Nov 30. PMID 27951433
- [Background] Alsawy S, Mansell W, McEvoy P, Tai S. What is good communication for people living with dementia? A mixed-methods systematic review. Int Psychogeriatr. 2017 Nov;29(11):1785-1800. doi: 10.1017/S1041610217001429. Epub 2017 Jul 31. PMID 28756788
- [Background] Sari YM, Burton E, Lee DA, Hill KD. Current physiotherapy practice on delivering treatments for older people with dementia in Indonesia: A cross-sectional study. Physiother Res Int. 2022 Jan;27(1):e1931. doi: 10.1002/pri.1931. Epub 2021 Nov 2. PMID 34727408
- [Background] Hoel V, Feunou CM, Wolf-Ostermann K. Technology-driven solutions to prompt conversation, aid communication and support interaction for people with dementia and their caregivers: a systematic literature review. BMC Geriatr. 2021 Mar 4;21(1):157. doi: 10.1186/s12877-021-02105-0. PMID 33663401
- [Background] American Geriatrics Society Expert Panel on Person-Centered Care. Person-Centered Care: A Definition and Essential Elements. J Am Geriatr Soc. 2016 Jan;64(1):15-8. doi: 10.1111/jgs.13866. Epub 2015 Dec 2. PMID 26626262
- [Background] BUTLER RN. The life review: an interpretation of reminiscence in the aged. Psychiatry. 1963 Feb;26:65-76. doi: 10.1080/00332747.1963.11023339. No abstract available. PMID 14017386
- [Background] McKeown J, Clarke A, Repper J. Life story work in health and social care: systematic literature review. J Adv Nurs. 2006 Jul;55(2):237-47. doi: 10.1111/j.1365-2648.2006.03897.x. PMID 16866815
- [Background] Woods B, O'Philbin L, Farrell EM, Spector AE, Orrell M. Reminiscence therapy for dementia. Cochrane Database Syst Rev. 2018 Mar 1;3(3):CD001120. doi: 10.1002/14651858.CD001120.pub3. PMID 29493789
- [Background] Zarit SH, Chiusano C, Harrison AS, Sewell L, Krause C, Liu Y. Rehabilitation of persons with dementia: using technology to improve participation. Aging Ment Health. 2021 Mar;25(3):543-550. doi: 10.1080/13607863.2020.1711864. Epub 2020 Jan 16. PMID 31941356
- [Background] Lazar A, Demiris G, Thompson HJ. Evaluation of a multifunctional technology system in a memory care unit: Opportunities for innovation in dementia care. Inform Health Soc Care. 2016 Dec;41(4):373-86. doi: 10.3109/17538157.2015.1064428. Epub 2016 Jan 28. PMID 26819070
- [Background] Cooney A, O'Shea E. The impact of life story work on person-centred care for people with dementia living in long-stay care settings in Ireland. Dementia (London). 2019 Oct-Nov;18(7-8):2731-2746. doi: 10.1177/1471301218756123. Epub 2018 Feb 7. No abstract available. PMID 29411663
- [Background] Rashid MH, Zahid MF, Zain S, Kabir A, Hassan SU. The Neuroprotective Effects of Exercise on Cognitive Decline: A Preventive Approach to Alzheimer Disease. Cureus. 2020 Feb 11;12(2):e6958. doi: 10.7759/cureus.6958. PMID 32190507
- [Background] Crocker T, Forster A, Young J, Brown L, Ozer S, Smith J, Green J, Hardy J, Burns E, Glidewell E, Greenwood DC. Physical rehabilitation for older people in long-term care. Cochrane Database Syst Rev. 2013 Feb 28;2013(2):CD004294. doi: 10.1002/14651858.CD004294.pub3. PMID 23450551
- [Background] Hall AJ, Burrows L, Lang IA, Endacott R, Goodwin VA. Are physiotherapists employing person-centred care for people with dementia? An exploratory qualitative study examining the experiences of people with dementia and their carers. BMC Geriatr. 2018 Mar 2;18(1):63. doi: 10.1186/s12877-018-0756-9. PMID 29499661
- [Background] Kales HC, Gitlin LN, Lyketsos CG; Detroit Expert Panel on Assessment and Management of Neuropsychiatric Symptoms of Dementia. Management of neuropsychiatric symptoms of dementia in clinical settings: recommendations from a multidisciplinary expert panel. J Am Geriatr Soc. 2014 Apr;62(4):762-9. doi: 10.1111/jgs.12730. Epub 2014 Mar 17. PMID 24635665
- [Background] Kitching D. Depression in dementia. Aust Prescr. 2015 Dec;38(6):209-2011. doi: 10.18773/austprescr.2015.071. Epub 2015 Dec 1. PMID 26843714
- [Background] Burks HB, des Bordes JKA, Chadha R, Holmes HM, Rianon NJ. Quality of Life Assessment in Older Adults with Dementia: A Systematic Review. Dement Geriatr Cogn Disord. 2021;50(2):103-110. doi: 10.1159/000515317. Epub 2021 Jun 24. PMID 34167127
- [Background] Creavin ST, Wisniewski S, Noel-Storr AH, Trevelyan CM, Hampton T, Rayment D, Thom VM, Nash KJ, Elhamoui H, Milligan R, Patel AS, Tsivos DV, Wing T, Phillips E, Kellman SM, Shackleton HL, Singleton GF, Neale BE, Watton ME, Cullum S. Mini-Mental State Examination (MMSE) for the detection of dementia in clinically unevaluated people aged 65 and over in community and primary care populations. Cochrane Database Syst Rev. 2016 Jan 13;2016(1):CD011145. doi: 10.1002/14651858.CD011145.pub2. PMID 26760674
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Lenze EJ, Munin MC, Quear T, Dew MA, Rogers JC, Begley AE, Reynolds CF 3rd. The Pittsburgh Rehabilitation Participation Scale: reliability and validity of a clinician-rated measure of participation in acute rehabilitation. Arch Phys Med Rehabil. 2004 Mar;85(3):380-4. doi: 10.1016/j.apmr.2003.06.001. PMID 15031821
- [Background] Weyer G, Erzigkeit H, Kanowski S, Ihl R, Hadler D. Alzheimer's Disease Assessment Scale: reliability and validity in a multicenter clinical trial. Int Psychogeriatr. 1997 Jun;9(2):123-38. doi: 10.1017/s1041610297004298. PMID 9309486
- [Background] Korner A, Lauritzen L, Abelskov K, Gulmann N, Marie Brodersen A, Wedervang-Jensen T, Marie Kjeldgaard K. The Geriatric Depression Scale and the Cornell Scale for Depression in Dementia. A validity study. Nord J Psychiatry. 2006;60(5):360-4. doi: 10.1080/08039480600937066. PMID 17050293
- [Background] Gbiri CAO, Amusa BF. Progressive task-oriented circuit training for cognition, physical functioning and societal participation in individuals with dementia. Physiother Res Int. 2020 Oct;25(4):e1866. doi: 10.1002/pri.1866. Epub 2020 Aug 10. PMID 32776698
- [Background] AsanoT, Wang C-W, Tsugaruva M, Ishikawa T. Effectiveness of high- frequency individual reminiscence interventions using life story books on person with dementia. British Journal of Occupational therapy. 2021:84(5):317-326.
- [Result] Duong S, Patel T, Chang F. Dementia: What pharmacists need to know. Can Pharm J (Ott). 2017 Feb 7;150(2):118-129. doi: 10.1177/1715163517690745. eCollection 2017 Mar-Apr. No abstract available. PMID 28405256
- [Result] Elfrink TR, Zuidema SU, Kunz M, Westerhof GJ. Life story books for people with dementia: a systematic review. Int Psychogeriatr. 2018 Dec;30(12):1797-1811. doi: 10.1017/S1041610218000376. Epub 2018 Jul 18. PMID 30017005
- See also: Life Story Questionnaire — http://www.crisisprevention.com/Blog/Use-This-Life-Story-Questionnaire-for-More-Person
- See also: Statistic software — http://www.gpower.hhu.de/
- See also: Statistic software — http://www.jamovi.org

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT05827276/Prot_SAP_ICF_001.pdf